CLINICAL TRIAL: NCT04532723
Title: Exoskeleton-Assisted Walking ExoAtlet II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company lost funding
Sponsor: Craig Hospital (Other)
Collaborators: COSMO ROBOTICS CO., Ltd (Industry)
Responsible Party: Principal Investigator, Candace Tefertiller, Executive Director of Research and Evaluation; PT,DPT,PhD,NCS, Craig Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRBNet ID 1559813
Record Dates: First submitted 2020-07-15; First posted 2020-08-31 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ExoAtlet II (Experimental): Safety/feasibility of utilizing the ExoAtlet II in a clinical setting with a group of individuals with SCI
  Interventions: Device: ExoAtlet II

INTERVENTIONS:
Device: ExoAtlet II — ExoAtlet II is the second version of an exoskeleton that ExoAtlet has manufactured

SUMMARY:
Based on prior exoskeleton research, it was determined that 40 participants of variable height, weight and injury level would provide a significant measure of the safety and feasibility of using the ExoAtlet II in individuals with SCI for standing and walking rehabilitation therapy. Craig Hospital will be responsible for enrolling up to 30 individuals during the study duration.The inclusion criteria will be utilized to identify appropriate subjects for this study.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord injury with lower extremity paralysis (partial or complete) levels T4-L5 (AIS A-C) or C7-T3 (AIS D)
* 18 Years of age or older in general good health
* Weight, no more than 220lbs (100kg)
* Intact Skin
* Able to stand without exhibiting symptomatic hypotension
* Use a wheelchair for mobility at least 50% of the day
* Enough strength in hands and shoulders to support standing and walking using crutches or a walker
* Medical clearance for full weight-bearing

  ---Per our clinical guidelines, we will require all individuals with SCI who are going to use an exoskeleton to receive full weight-bearing medical clearance from their physician prior to participation. If they are unable to obtain full weight-bearing medical clearance they will not be able to participate in this study.
* Passive range of motion (PROM) at shoulders, trunk, upper extremities and lower extremities within functional limits for safe gait and use of appropriate assistive device/stability aid
* Hip width no greater than 18" (46 cm) measured when sitting
* Femur length between 37 cm and 49 cm measured between mid-patellar tendon and the floor

Exclusion Criteria:

* Spinal cord injury level higher than T4 (AIS A-C) or C7 ASIA D
* Severe muscle stiffness/tightness
* Significant spasticity (Modified Ashworth Scale score of 3 or above)
* Trunk or lower extremity pressure wound
* Unstable spine, un-healed limbs, or fractures
* Presence of bone in soft tissue where bone normally does not exist (heterotopic ossification), limiting range of motion in the hip or knee joints

  ---Each individual who is interested in participating in this study will be screened for heterotropic ossification (HO) using a verbal checklist first and then they participate in a thorough range of motion (ROM) evaluation before being fit in the exoskeleton. If they verbalize a history of HO or demonstrate a bony block/resistance to passive ROM, they will be sent back to their physician to rule out HO and will not participate in the study until they receive additional clearance.
* Joint instability, dislocation, moderate to severe hip dysplasia
* Uncontrolled seizures
* Fracture or lower-limb surgery in past year
* Psychopathology, or other condition that the physician or investigator, in his or her clinical judgment, considers to be exclusionary to safely use an exoskeleton
* Pregnant or lactating females (Potential female participants will be informed that risks to pregnant or lactating females are unknown; then they will be asked if they are pregnant or lactating, or if they could be pregnant. If there is any uncertainty, they will not be included in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Integrity | change from baseline skin integrity at 2 weeks
  Skin breakdown
Change in Falls | change from baseline number of falls at 2 weeks
  Number of falls
Change in Fractures | change from baseline number of fractures at 2 weeks
  Number of fractures and cause

SECONDARY OUTCOMES:
Heart Rate | Baseline, Week 1
  Heart rate beats per minute
Blood pressure | Baseline, Week 1
  Blood pressures mm/Hg
Spasticity | Baseline, Week 1, Week 2
  Modified Ashworth
Standing Time | Baseline, Week 1
  Upright and weight bearing total time
Ambulation Time | Week 1
  Total walking time
Standing Assistance | Baseline, Week 1
  level of assistance in standing
Ambulation Assistance | Week 1
  Level of assistance for walking
6 Minute Walk Test | Week 1
  Total distance walked in 6 minutes
10 Meter Walk Test | Week 1
  total time to walk 10 meters
Physical Activity Enjoyment Scale | Baseline, Week 1, Week 2
  Scale of participant enjoyment in the moment. 7-point bipolar rating scale, eleven items are reverse scored. Higher total score reflect greater levels of enjoyment
BORG Rate of Perceived Exertion | Baseline, Week 1
  Scale of participant effort. Lowest score is 6 and 20 is highest score. Higher scores reflect greater effort exerted by participant